CLINICAL TRIAL: NCT05381441
Title: A Cluster Randomized Controlled Trial Comparing the Safety Action Feedback and Engagement (SAFE) Loop With an Established Incident Reporting System
Brief Title: Safety Action Feedback and Engagement (SAFE) Loop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Teryl K. Nuckols, Vice Chair for Clinical Research, Director of Division of General Internal Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00001025; R01HS027455 (AHRQ)
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Medication Errors; Patient Safety
Keywords: Incident Reporting; Implementation Sciences; Nursing Research; Risk Management; Hospital

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial randomizing blocks of nursing units to either the control or intervention group
Who Masked: Participant, Outcomes Assessor
Masking Description: Nurses and nursing units will not be masked to study arm. Patients cared for on nursing units will be masked to study arm (and will not be consented for participation). Outcome assessors will be blinded to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE Loop Arm (Experimental): Nursing units involved in the intervention arm will participate in an iterative educational and quality improvement process that encourages improved reporting of medication safety events deemed important to their individual nursing units.
  Interventions: Behavioral: Safety Action Feedback and Engagement (SAFE) Loop
- Control Arm (No Intervention): Nurses in this study will continue standard practice protocol.

INTERVENTIONS:
Behavioral: Safety Action Feedback and Engagement (SAFE) Loop — Nursing units randomized to the intervention arm will undergo the SAFE Loop intervention, which involves five Key Attributes: (1) obtaining input from nurses on which problems to address; (2) focusing on selected high-priority events, (3) prompting nurses to report the high-priority events for a designated period and write more informative reports; (4) following standardized investigative procedures to integrate information from sources internal and external to CSMC, and (5) providing feedback to nurses about safety problems and mitigation plans. During all phases, the SAFE Loop Team collaborates with frontline nurses and Unit Managers.
  Arms: SAFE Loop Arm

SUMMARY:
This trial will test whether a new intervention, the Safety Action Feedback and Engagement (SAFE) Loop, enhances nurse incident reporting practices, improves nurses' perceptions of incident reporting, and lowers rates of high-priority medication events, as compared with using an existing incident reporting system. The trial will be performed in 20 acute care nursing units at Cedars-Sinai Medical Center.

DETAILED DESCRIPTION:
This cluster randomized controlled trial will test whether a novel intervention, the Safety Action Feedback and Engagement (SAFE) Loop, enhances hospital incident reporting practices, improves nurses' perceptions of incident reporting, and lowers rates of high-priority medication events, as compared with Cedars-Sinai Medical Center's (CSMC's) existing incident reporting system.

The specific aims are to determine whether SAFE Loop:

* Aim 1: improves incident reporting practices by increasing the rate at which nurses report high-priority medication incidents (H1.1) and the number of contributing factors described per report (H1.2).
* Aim 2: improves nurses' attitudes toward incident reporting, including perceptions of feedback and communication about error (H2.1) and of the frequency with which events are reported (H2.2).
* Aim 3: reduces rates of high-priority medication events (H3.1) and high-priority medication events involving harm (H3.2).

Setting and Subject Population: 20 acute care nursing units at Cedars-Sinai Medical Center in Los Angeles, where about 1980 nurses provide over 294,000 patient-days of care per year (about 115,000 hospital visits).

Quality Improvement (QI) Activities: (1) Safe Loop Activities, including obtaining input from nurses, educational activities training them in how to focus on target events and write high-quality reports, stimulated time-limited reporting, integration of information from reports and other QI data sources from within the hospital and other information, designing changes to improve medication safety, and providing feedback to nurses. (2) Randomization of nursing units to intervention or control and early vs. later implementation. The will assure that the implementation occurs in a uniform and manageable fashion. (3) Implementation activities: planning, engaging, executing, reflecting/evaluating.

Primary Research Procedures:

1. Nurse surveys (N=1,980): We will attempt to survey about 1980 nurses on study nursing units. Survey recruitment will be done through email, with e-informed consent via Redcap.
2. Nurse interviews on implementation (N=37): We will interview 32 nurses (10 unit leaders and 22 registered nurses) to characterize implementation. We will recruit nurses and unit leaders will by email and word-of-mouth. Prelim work: We will conduct cognitive tests of the interview script with up to 5 nurses to make refinements (2 unit leaders, 3 floor nurses)
3. Analysis of Incident Reports (N=1,963): We will examine incident reports related to medication events during the study period. We anticipate that 1,663 patients will have eligible incident reports. Prelim work: We will conduct practice analyses on up to 300 patients with incident reports to refine study instruments and train analysts. We may seek to publish findings based on prelim work.
4. Analysis of Medication Events (N=1,520): We will randomly sample 1,520 hospitalizations during the study period. We will review medical records and access pharmacy iVents reports to identify events. We will also obtain variables from the electronic health record on all these patients as well (for case mix adjustment). Prelim work: We will conduct practice analyses on up to 100 medical records to refine instruments and train nurse and physician analysts.
5. Nurse interviews for DSM (N=18): As part of our Data Safety and Monitoring Plan, we will interview 15 nurses on the intervention nursing units that first implement the intervention to assess and monitor for adverse consequences to the nurses. We will recruit nurses by having a research nurse go to the nursing units and ask to speak with nurses privately. Preliminary work: We will pilot test the interview guide with 3-5 nurses.

Total number of hospital visits: Approximately 172,500 over 2.5 years. Length of follow up: start of hospital visit (e.g., admission) to discharge from hospital or end of study, whichever is earlier.

How Participation Differs from Standard of Care: In current systems of hospital care, voluntary incident reporting is a technique through which frontline personnel -usually nurses-submit reports that describe events that posed risks to safety, particularly incidents that were intercepted or happened not to cause harm. In contrast, participation in the study involves the Safety Action Feedback and Engagement (SAFE) Loop. The SAFE Loop has five key attributes designed to transform hospital incident reporting systems into much more effective tools for improving patient safety: obtaining nurses' input about which medication safety problems to address; focusing on selected high-priority medication events; prompting nurses to report high-priority medication events during a designated period and training them to write more informative reports; integrating information about medication safety problems on hospital nursing units from the incident reports, investigations, and other internal and external sources; and providing feedback to nurses on the problems identified on the nursing units and mitigation plans.

Any parts of the protocol not conducted at CSMC? Not applicable. All parts will be conducted at CSMC.

Advancing knowledge or clinical practice: This study will be a highly rigorous and comprehensive evaluation of an incident reporting intervention in healthcare. This appears to be the first RCT of an intervention designed to improve incident reporting in healthcare, and the first study to examine the effect of an incident reporting intervention on an important patient safety outcome, medication event rates. Prior studies have only used observational designs and examined effects on the timeliness of reporting, the numbers of reports, and the types of incidents reported.

Lastly, this study will transform how incident reporting systems function in hospitals: (A) Engaging Nurses in Decisions about Which Patient Safety Problems to Address. Prior strategies for improving safety include top-down initiatives. However, clinician engagement is essential because safety is an emergent property that results from millions of small actions they take each day. (B) Prompting Nurses to Report High-priority Events and Write More Informative Reports. Emphasizing high-priority events increases the likelihood of making meaningful improvements in safety. This project emphasizes the value of incident reporting as a tool for gaining insights into the causes of critical events, based on successes of incident reporting at improving safety in other high-risk industries. (C) Creating Standardized Procedures for Investigating High-priority Events. Procedures for following up on reports are variable and not well standardized; therefore, this will be a major advance in the field. (D) Providing Feedback to Nurses about How Reports Were Used to Improve Safety. Interventions that improve incident reporting are more likely to succeed and be sustained if frontline clinicians receive feedback that their reports were useful and observe changes in systems of care and event rates-experts call this the 'safety action feedback loop.' Few interventions have attempted to strengthen this loop in healthcare.

ELIGIBILITY:
Nurses:

Inclusion Criteria:

1. Intervention (SAFE Loop):

   * All 1,980 nurses on the nursing units will be eligible to participate.
2. Aim 1 (review of incident reports):

   * All 1,980 nurses on the nursing units will be eligible to participate.
3. Aim 2 (survey of nurses):

   * Nurses will be eligible if they worked >50% time on one study nursing unit during a 6-month study period.
4. Aim 3 (review of medical records):

   * All 1,980 nurses on the nursing units will be eligible to participate.
5. Qualitative interviews:

   * Nurses and nurse managers will be eligible to participate if they worked at least 50% time on the study nursing units for the entire duration of a SAFE Loop implementation period.
   * We will enroll 32 participants out of a pool of approximately 800 eligible nurses.

Exclusion Criteria:

1. All study procedures:

   * Provided care ONLY in outpatient clinics, operating/ procedure rooms, post-anesthesia care, and diagnostic and therapeutic services.
2. Aim 3:

   * Provided care ONLY in the emergency department.

Patients:

Inclusion Criteria:

1. Intervention (SAFE Loop):

   * All patients admitted to the study nursing units during a 6-month study period will be eligible to participate.
2. Aim 1 (review of incident reports):

   * Patients will be cared for on the study nursing units during a 6-month study period.
   * Patients will also have an incident report that addresses one of the high-priority medication events.
3. Aim 2 (survey of nurses):

   * Not applicable.
4. Aim 3 (review of medical records):

   * Patients will be admitted to the study nursing units during a 6-month study period.
   * We will randomly sample 1,520 hospitalizations divided equally between the four study groups and the baseline and follow-on periods.
5. Qualitative interviews:

   * Not applicable.

Exclusion Criteria:

1. All study procedures:

   * Received care ONLY in outpatient clinics, operating/ procedure rooms, post-anesthesia care, and diagnostic and therapeutic services.
2. Aim 3:

   * Received care ONLY in the emergency department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5163 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Nurses' incident reporting practices | 48 weeks
  Number of work-system factors identifiable in the narrative section of each incident report. Two researchers with expertise in human factors methods will identify (and classify) the work-system factors described in each incident report, with a third researcher available to adjudicate ties. Work-system factors will be based on HFACS Healthcare taxonomy.
Nurses' attitudes regarding communication about error | 24 weeks
  Performance on composite measure on "Communication About Error," from AHRQ Hospital Survey on Patient Safety Culture™ version 2.0, based on surveys of nurses.
Rate of high-priority medication events | 48 weeks
  Rate per 1,000 patient-days of medication events identified as high priorities for prevention by the 10 nursing units in the intervention group. Medication events include preventable adverse drug events and potential adverse drug events. Medication events will be detected via the IHI Trigger Tool method of medical record review, with screening by trained nurse reviewers and confirmation by trained physician reviewers.

SECONDARY OUTCOMES:
Rate of reporting high-priority medication events | 48 weeks
  Rate (%) per 1000 patient-days of incident reports addressing one of the medication events identified as high priorities for prevention by the 10 nursing units in the intervention group. Medication events include preventable adverse drug events and potential adverse drug events.
Nurses' attitudes regarding reporting of patient safety events | 24 weeks
  Performance on composite measure on "Reporting Patient Safety Events," from AHRQ Hospital Survey on Patient Safety Culture™ version 2.0, based on surveys of nurses.
Rate of high-priority medication events that involved patient harm | 48 weeks
  Rate per 1,000 patient-days of medication events (1) identified as high priorities for prevention by the 10 nursing units in the intervention group, and (2) involving harm (NCC MERP severity categories E-I). These medication events will include only preventable adverse drug events (NOT potential adverse drug events). Medication events will be detected via the IHI Trigger Tool method of medical record review, with screening by trained nurse reviewers and confirmation and classification (severity rating) by trained physician reviewers.

CONTACTS AND LOCATIONS:
Overall Officials: Teryl K Nuckols, MD, Principal Investigator — Vice Chair for Clinical Research Dept of Medicine, Cedars-Sinai; Carl Berdahl, MD, Study Director — Physician Scientist, Cedars-Sinai
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen TN, Francis SE, Wiegmann DA, Shappell SA, Gewertz BL. Using HFACS-Healthcare to Identify Systemic Vulnerabilities During Surgery. Am J Med Qual. 2018 Nov/Dec;33(6):614-622. doi: 10.1177/1062860618764316. Epub 2018 Mar 21. PMID 29562768
- [Derived] Seferian E, Berdahl CT, Coleman B, Leang D, Cohen T, Qureshi N, McCleskey SG, Kaiser K, Grissinger M, Kanji F, Henreid AJ, Carrascoza-Bolanos J, Daniels L, Abarca O Jr, De La Cruz P, Truong BT, Nuckols TK. The Safety Action Feedback and Engagement (SAFE) Loop: Initial Testing and Refinement of a Novel Intervention to Enhance Hospital Incident Reporting and Patient Safety. medRxiv [Preprint]. 2025 Jun 6:2025.06.03.25328744. doi: 10.1101/2025.06.03.25328744. PMID 40502590
- See also: IHI Trigger Tool Method — http://www.ihi.org/resources/Pages/Tools/IHIGlobalTriggerToolforMeasuringAEs.aspx
- See also: NCC MERP Classification of Medication Errors — https://www.nccmerp.org/categorizing-medication-errors-index-color
- See also: AHRQ Hospital Survey on Patient Safety Culture version 2 — https://www.ahrq.gov/sops/surveys/hospital/index.html
- See also: HFACS Healthcare — https://hfacs-healthcare.com/

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT05381441/Prot_SAP_000.pdf
  • Informed Consent Form: Nurse Surveys (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05381441/ICF_001.pdf
  • Informed Consent Form: Nurse Interviews (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05381441/ICF_002.pdf